CLINICAL TRIAL: NCT04605978
Title: A Phase IIa Efficacy and Safety Trial With Intravenous S95011 in Primary Sjögren's Syndrome Patients: An International, Multicentre, Randomised, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of S95011 in Primary Sjögren's Syndrome Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL2-95011-001; 2020-001526-59 (EudraCT Number)
Record Dates: First submitted 2020-10-19; First posted 2020-10-28 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Primary Sjögren's Syndrome
Keywords: Sjögren; Sjögren's Syndrome; Autoimmune disease; Systemic; Xerostomia; xerophthalmia; Salivary gland disease; Arthritis; Joint disease; Monoclonal antibody
MeSH Terms: conditions — Sjogren's Syndrome; Autoimmune Diseases; Xerostomia; Xerophthalmia; Salivary Gland Diseases; Arthritis; Joint Diseases | interventions — Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S95011 concentrate for solution for infusion (Experimental): S95011 is administrated by one IV infusion every 2 weeks for the first month and then every 3 weeks.
  Interventions: Drug: S95011 concentrate for solution for infusion
- S95011 Placebo concentrate for solution for infusion (Placebo Comparator): S95011 placebo is administrated by one IV infusion every 2 weeks for the first month and then every 3 weeks.
  Interventions: Drug: Placebo concentrate for solution for infusion

INTERVENTIONS:
Drug: S95011 concentrate for solution for infusion — IV administration every 2 weeks until week 4 and then every 3 weeks until week 10.
  Arms: S95011 concentrate for solution for infusion
Drug: Placebo concentrate for solution for infusion — IV administration every 2 weeks until week 4 and then every 3 weeks until week 10.
  Arms: S95011 Placebo concentrate for solution for infusion

SUMMARY:
The purpose of this study is to assess the effect of multiple intravenous infusions of S95011 compared to placebo in reducing disease activity in patients with primary Sjögren's syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary Sjögren's Syndrome based on 2016 American College of Rheumatology-EULAR criteria
2. ESSDAI total score ≥ 6 during screening, with at least 6 points scored within the 7 following domains: constitutional, lymphadenopathy, glandular, articular, cutaneous, hematologic and biologic,
3. Positive anti-Sjögren's Syndrome A (Ro) antibodies or anti-nuclear antibodies (ANA) ≥ 1:320 or rheumatoid factor (RF) >20 IU/ml during screening period, measured in a central laboratory
4. Stimulated whole salivary flow rate > 0 mL/minute

Exclusion Criteria:

1. Prior administration within the timeframe described in the protocol of any of the following:

   * Belimumab,
   * Rituximab or other B cell depleting agents,
   * Abatacept,
   * Tumor necrosis factor inhibitors,
   * Tocilizumab,
   * Cyclophosphamide,
   * Cyclosporine (except for eye drops), tacrolimus, sirolimus, mycophenolate mofetil (MMF), azathioprine, or leflunomide
   * Janus kinase (JAK) inhibitors
2. Meeting any of the following conditions:

   * Corticosteroids: > 10 mg/day oral prednisone (or equivalent) within 4 weeks prior to randomisation (W000); Any change or initiation of new dose of oral prednisone (or equivalent) within 4 weeks prior to randomisation (W000); Intramuscular, IV, or intra-articular corticosteroids within 4 weeks prior to randomisation (W000); Any change or initiation of new dose of topical corticosteroids within 2 weeks prior to randomisation (W000),
   * Antimalarials: any change or initiation of new dose of antimalarials (e.g. chloroquine, hydroxychloroquine, quinacrine) within 16 weeks prior to randomisation (W000),
   * Methotrexate: > 25 mg/week of methotrexate; any initiation or change of dose of methotrexate within 12 weeks prior to randomisation (W000); any change in route of administration within 4 weeks prior to randomisation (W000),
   * Non-steroidal anti-inflammatory drugs (NSAIDs): Any change or initiation of new dose of regularly scheduled NSAIDs within 2 weeks prior to randomisation (W000),
   * Cevimeline or pilocarpine and cyclosporine eye drops (Restasis) and lifitegrast: any increase or initiation of new doses within 2 weeks prior to randomisation (W000).
3. Secondary Sjögren's Syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (2):
  - Colorado Arthritis Associates, Lakewood, Colorado
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
- The Queen Elizabeth Hospital Rheumatology Unit, Woodville, Australia
- France (5):
  - Hôpital Saint-André, Bordeaux
  - CHU de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Laribiosière, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris
- Germany (2):
  - Universitätsklinikum Erlangen Medizinische Klinik 3 Rheumatologie und Immunologie, Erlangen
  - Universitätsklinikum Freiburg Department Innere Medizin Klinik für Rheumatologie und Klinische Immunologie, Freiburg im Breisgau
- Hungary (3):
  - Debreceni Egyetem Orvos és Egészségtudományi Centrum Belgyógyászat C épület - Klinikai Immunológiai Tanszék, Debrecen
  - Békés Megyei Központi Kórház, Pándy Kálmán Tagkórház, Infektológia-Hepatológia, Gyula
  - Vita Verum Medical Bt. Berényi u. 72-100. 95. számú épület 16. Rendelő, Székesfehérvár
- Spain (3):
  - CLINICA SAGRADA FAMILIA Servicio de Reumatología y Unidad de Ensayos Clínicos, Barcelona
  - CLINICAL GAIAS SANTIAGO Servicio de Reumatología, Santiago de Compostela
  - Hospital Infanta Luisa Quirón Salud Servicio de Reumatología, Seville
- United Kingdom (3):
  - Queen Elizabeth Hospital, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Freeman Hospital, Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Southampton General Hospital, University Hospital Southampton NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH).
  The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- See also: Find Results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- S95011 Concentrate for Solution for Infusion: S95011 was administrated by one IV infusion every 2 weeks for the first month and then every 3 weeks.
- S95011 Placebo Concentrate for Solution for Infusion: S95011 placebo was administrated by one IV infusion every 2 weeks for the first month and then every 3 weeks.
Period: Overall Study
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion
Started | 31 | 17
Completed | 28 | 15
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal nonmedical reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion | Total
Number analyzed (Participants) | 31 | 17 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (12.6) | 53.6 (12.5) | 53.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 16 | 42
  Male | 5 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 28 | 16 | 44
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 2 | 0 | 2
  Race: Black or African American | 1 | 0 | 1
  Race: Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Race: Other | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1 | 1 | 2
  Ethnicity: Not Hispanic or Latino | 30 | 16 | 46
Duration since diagnosis of pSS (years) [Mean (Standard Deviation); unit: years] | 7.6 (7.7) | 6.5 (6.6) | 7.2 (7.3)
Patient taking a specific treatment for pSS (for randomization stratification) [Count of Participants; unit: Participants]
  Nothing | 17 | 8 | 25
  Oral corticosteroid | 4 | 1 | 5
  Antimalarial | 5 | 5 | 10
  Oral corticosteroid and antimalarial | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in ESSDAI Total Score
Description: Efficacy criterion Eular Sjögren Syndrome Disease Activity index (ESSDAI) is a physician-administered clinical index which has been validated to objectively assess systemic manifestations in Primary Sjögren's Syndrome patients. Scores range from 0 - 123, with a lower score representing less disease activity.
Time Frame: From baseline to week 13
Population: Change in ESSDAI Total Score is computed only on observed values before occurrence of Intercurrent Events.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion
Number analyzed (Participants) | 31 | 17
score on a scale
  Change from Baseline to Week 13: number analyzed (Participants) | 26 | 13
  Change from Baseline to Week 13 | -3.77 (4.55) | -5.54 (4.89)
  Baseline | 11.52 (3.75) | 13.12 (7.20)
  Week 13: number analyzed (Participants) | 26 | 13
  Week 13 | 7.96 (4.91) | 8.85 (8.59)
Statistical Analysis 1: Comparison: S95011 Concentrate for Solution for Infusion; Test type: Superiority; Mean Difference (Net) = 2.44, 95% CI 2-sided [-0.61 to 5.49] — Missing data and data post intercurrent event were imputed for the statistical analysis as specified in the statistical analysis plan

2. Secondary Outcome: ESSDAI Score by Domain and Total Score
Description: Efficacy criterion Eular Sjögren Syndrome Disease Activity index (ESSDAI) is a physician-administered clinical index which has been validated to objectively assess systemic manifestations in Primary Sjögren's Syndrome patients. There are 12 organ-specific domains and for each domain, features of disease activity are scored according to their severity. These scores are then summed across the 12 domains in a weighted manner to provide the total score. The total score ranges from 0 to 123. A higher score always represents a more severe disease activity. The domain [weight] and score range are as follows: Constitutional [3] 0-2; Lymphadenopathy and lymphoma [4] 0-3; Glandular [2] 0-2; Articular [2] 0-3; Cutaneous [3] 0-3; Pulmonary [5] 0-3; Renal [5] 0-3; Muscular [6] 0-3; PNS [5] 0-3; CNS [5] 0-3; Hematological [2] 0-3; Biological [1] 0-2.
Time Frame: At baseline, week 4 and week 13
Population: ESSDAI Score by Domain and Total Score is computed without consideration of Intercurrent Events, therefore data gathered after an intercurrent event is not set as "missing". The participant data that is missing from Week 4 and Week 13 was not available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion
Number analyzed (Participants) | 31 | 17
score on a scale
  Total Score - Baseline | 11.5 (3.7) | 13.1 (7.2)
  Total Score - Week 4: number analyzed (Participants) | 31 | 16
  Total Score - Week 4 | 9.5 (3.7) | 10.8 (7.2)
  Total Score - Week 13: number analyzed (Participants) | 28 | 15
  Total Score - Week 13 | 7.8 (4.8) | 9.7 (8.3)
  Constitutional - Baseline | 0.6 (0.7) | 0.4 (0.6)
  Constitutional - Week 4: number analyzed (Participants) | 31 | 16
  Constitutional - Week 4 | 0.5 (0.7) | 0.2 (0.4)
  Constitutional - Week 13: number analyzed (Participants) | 28 | 15
  Constitutional - Week 13 | 0.4 (0.7) | 0.2 (0.6)
  Lymphadenopathy and lymphoma - Baseline | 0.5 (0.8) | 0.6 (0.6)
  Lymphadenopathy and lymphoma - Week 4: number analyzed (Participants) | 31 | 16
  Lymphadenopathy and lymphoma - Week 4 | 0.3 (0.7) | 0.3 (0.5)
  Lymphadenopathy and lymphoma - Week 13: number analyzed (Participants) | 28 | 15
  Lymphadenopathy and lymphoma - Week 13 | 0.4 (0.7) | 0.4 (0.5)
  Glandular - Baseline | 0.7 (0.7) | 0.7 (0.7)
  Glandular - Week 4: number analyzed (Participants) | 31 | 16
  Glandular - Week 4 | 0.6 (0.6) | 0.6 (0.6)
  Glandular - Week 13: number analyzed (Participants) | 28 | 15
  Glandular - Week 13 | 0.4 (0.6) | 0.5 (0.7)
  Articular - Baseline | 1.5 (1.1) | 1.6 (1.2)
  Articular - Week 4: number analyzed (Participants) | 31 | 16
  Articular - Week 4 | 1.1 (1.1) | 1.3 (1.3)
  Articular - Week 13: number analyzed (Participants) | 28 | 15
  Articular - Week 13 | 0.6 (0.7) | 0.7 (1.0)
  Cutaneous - Baseline | 0.3 (0.6) | 0.1 (0.5)
  Cutaneous - Week 4: number analyzed (Participants) | 31 | 16
  Cutaneous - Week 4 | 0.2 (0.6) | 0.1 (0.5)
  Cutaneous - Week 13: number analyzed (Participants) | 28 | 15
  Cutaneous - Week 13 | 0.3 (0.6) | 0.2 (0.8)
  Pulmonary - Baseline | 0.0 (0.2) | 0.3 (0.6)
  Pulmonary - Week 4: number analyzed (Participants) | 31 | 16
  Pulmonary - Week 4 | 0.0 (0.2) | 0.3 (0.6)
  Pulmonary - Week 13: number analyzed (Participants) | 28 | 15
  Pulmonary - Week 13 | 0.0 (0.0) | 0.2 (0.6)
  Renal - Baseline | 0.0 (0.0) | 0.0 (0.0)
  Renal - Week 4: number analyzed (Participants) | 31 | 16
  Renal - Week 4 | 0.0 (0.0) | 0.0 (0.0)
  Renal - Week 13: number analyzed (Participants) | 28 | 15
  Renal - Week 13 | 0.0 (0.0) | 0.0 (0.0)
  Muscular - Baseline | 0.0 (0.0) | 0.0 (0.0)
  Muscular - Week 4: number analyzed (Participants) | 31 | 16
  Muscular - Week 4 | 0.0 (0.0) | 0.0 (0.0)
  Muscular - Week 13: number analyzed (Participants) | 28 | 15
  Muscular - Week 13 | 0.0 (0.0) | 0.0 (0.0)
  Peripheral Nervous System (PNS) - Baseline | 0.1 (0.2) | 0.2 (0.5)
  Peripheral Nervous System (PNS) - Week 4: number analyzed (Participants) | 31 | 16
  Peripheral Nervous System (PNS) - Week 4 | 0.0 (0.2) | 0.2 (0.5)
  Peripheral Nervous System (PNS) - Week 13: number analyzed (Participants) | 28 | 15
  Peripheral Nervous System (PNS) - Week 13 | 0.0 (0.2) | 0.2 (0.6)
  Central Nervous System (CNS) - Baseline | 0.0 (0.0) | 0.1 (0.5)
  Central Nervous System (CNS) - Week 4: number analyzed (Participants) | 31 | 16
  Central Nervous System (CNS) - Week 4 | 0.0 (0.0) | 0.1 (0.5)
  Central Nervous System (CNS) - Week 13: number analyzed (Participants) | 28 | 15
  Central Nervous System (CNS) - Week 13 | 0.0 (0.0) | 0.1 (0.5)
  Hematological - Baseline | 0.6 (0.7) | 0.4 (0.5)
  Hematological - Week 4: number analyzed (Participants) | 31 | 16
  Hematological - Week 4 | 0.7 (0.7) | 0.5 (0.5)
  Hematological - Week 13: number analyzed (Participants) | 28 | 15
  Hematological - Week 13 | 0.8 (0.8) | 0.4 (0.5)
  Biological - Baseline | 0.9 (0.8) | 0.8 (0.8)
  Biological - Week 4: number analyzed (Participants) | 31 | 16
  Biological - Week 4 | 0.9 (0.8) | 0.9 (0.9)
  Biological - Week 13: number analyzed (Participants) | 28 | 15
  Biological - Week 13 | 0.8 (0.8) | 1.1 (0.9)

3. Secondary Outcome: ESSPRI Score by Symptom and Total Score
Description: Efficacy criterion EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) is an index designed to measure patients' symptoms in primary Sjögren's Syndrome. The three domains included in this scale are dryness, fatigue, and pain, each of which are scored on a scale of 0-10. The total score is calculated as the average of the three domain scores and therefore the maximum total score is 10. The higher score represents more severe symptoms.
Time Frame: At baseline, week 4 and week 13
Population: The number of analyzed participants at each timepoint is different than the overall number of participants analyzed due to missing data (e.g. some participants have missing data at baseline but observed data at other timepoints and inversely)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion
Number analyzed (Participants) | 31 | 17
score on a scale
  Total score - Baseline: number analyzed (Participants) | 28 | 17
  Total score - Baseline | 7.14 (1.59) | 6.87 (1.65)
  Total score - Week 4: number analyzed (Participants) | 24 | 14
  Total score - Week 4 | 6.65 (1.83) | 5.19 (1.97)
  Total score - Week 13: number analyzed (Participants) | 24 | 13
  Total score - Week 13 | 5.54 (2.06) | 5.40 (2.71)
  Dryness score - Baseline: number analyzed (Participants) | 28 | 17
  Dryness score - Baseline | 7.46 (1.69) | 7.06 (2.38)
  Dryness score - Week 4: number analyzed (Participants) | 24 | 14
  Dryness score - Week 4 | 6.96 (2.20) | 5.64 (2.47)
  Dryness score - Week 13: number analyzed (Participants) | 24 | 13
  Dryness score - Week 13 | 6.54 (1.91) | 6.62 (2.43)
  Fatigue score - Baseline: number analyzed (Participants) | 28 | 17
  Fatigue score - Baseline | 7.43 (1.43) | 7.18 (2.24)
  Fatigue score - Week 4: number analyzed (Participants) | 24 | 14
  Fatigue score - Week 4 | 6.88 (2.15) | 5.29 (2.58)
  Fatigue score - Week 13: number analyzed (Participants) | 24 | 13
  Fatigue score - Week 13 | 5.71 (2.74) | 5.15 (3.21)
  Pain score - Baseline: number analyzed (Participants) | 28 | 17
  Pain score - Baseline | 6.54 (2.63) | 6.35 (2.21)
  Pain score - Week 4: number analyzed (Participants) | 24 | 14
  Pain score - Week 4 | 6.13 (2.85) | 4.64 (2.71)
  Pain score - Week 13: number analyzed (Participants) | 24 | 13
  Pain score - Week 13 | 4.38 (3.21) | 4.46 (3.57)

4. Secondary Outcome: Quality of Life (SF-36)
Description: Efficacy criterion The Short Form (SF-36) Health Survey is a 36-item, patient-reported survey of patient health to asses QoL. Scores for each subscale range from 0 - 100, with a lower number representing a worse quality of life.
Time Frame: At baseline and week 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion
Number analyzed (Participants) | 31 | 17
score on a scale
  Physical score - Baseline: number analyzed (Participants) | 28 | 17
  Physical score - Baseline | 38.729 (9.742) | 40.295 (8.236)
  Physical score - Week 13: number analyzed (Participants) | 23 | 13
  Physical score - Week 13 | 45.139 (9.409) | 47.011 (9.819)
  Mental score - Baseline: number analyzed (Participants) | 28 | 17
  Mental score - Baseline | 40.911 (10.909) | 44.182 (13.208)
  Mental score - Week 13: number analyzed (Participants) | 23 | 13
  Mental score - Week 13 | 41.970 (14.562) | 45.050 (14.275)

5. Secondary Outcome: Fatigue (MFI)
Description: Efficacy criterion Modified Fatigue Impact Scale (MFI) is a 20-item survey to evaluate ﬁve dimensions of fatigue. Scores range from 4 to 20 for each sub-score, with a lower score representing less fatigue.
Time Frame: At baseline and week 13
Population: The number of analyzed participants at each timepoint is different than the overall number of participants analyzed due to missing data (e.g. some participants have missing data at baseline (for all domains) but observed data at other timepoints and inversely).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion
Number analyzed (Participants) | 31 | 17
score on a scale
  General fatigue score - Baseline: number analyzed (Participants) | 28 | 17
  General fatigue score - Baseline | 15.1 (3.0) | 15.2 (3.6)
  General fatigue score - Week 13: number analyzed (Participants) | 23 | 13
  General fatigue score - Week 13 | 13.2 (3.5) | 13.5 (5.3)
  Physical fatigue score - Baseline: number analyzed (Participants) | 28 | 17
  Physical fatigue score - Baseline | 14.3 (2.7) | 13.9 (3.9)
  Physical fatigue score - Week 13: number analyzed (Participants) | 23 | 13
  Physical fatigue score - Week 13 | 12.6 (3.9) | 11.4 (5.2)
  Reduced activity score - Baseline: number analyzed (Participants) | 28 | 17
  Reduced activity score - Baseline | 12.9 (3.0) | 12.3 (3.8)
  Reduced activity score - Week 13: number analyzed (Participants) | 23 | 13
  Reduced activity score - Week 13 | 11.4 (4.7) | 9.7 (4.3)
  Reduced motivation score - Baseline: number analyzed (Participants) | 27 | 16
  Reduced motivation score - Baseline | 11.3 (4.1) | 9.1 (3.1)
  Reduced motivation score - Week 13: number analyzed (Participants) | 23 | 13
  Reduced motivation score - Week 13 | 10.3 (4.5) | 8.8 (4.5)
  Mental fatigue score - Baseline: number analyzed (Participants) | 28 | 17
  Mental fatigue score - Baseline | 11.6 (3.9) | 10.5 (3.7)
  Mental fatigue score - Week 13: number analyzed (Participants) | 23 | 13
  Mental fatigue score - Week 13 | 11.4 (4.9) | 9.5 (4.1)

6. Secondary Outcome: Physician's Global Assessment (PhGA) of the Disease Activity
Description: Efficacy criterion Physician's global assessment (PhGA) of the disease activity is a 0 to 10 numerical rating scale (NRS), with a lower score representing less disease activity.
Time Frame: At baseline and week 13
Population: The number analyzed for Week 13 is less due to missing patient data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion
Number analyzed (Participants) | 31 | 17
score on a scale
  Baseline | 6.0 (1.5) | 6.3 (1.3)
  Week 13: number analyzed (Participants) | 24 | 15
  Week 13 | 3.6 (1.3) | 4.2 (1.6)

7. Secondary Outcome: Patient's Global Assessment (PGA) of the Disease Activity
Description: Efficacy criterion Patient's global assessment (PGA) of the disease activity is a 0 to 10 numerical rating scale (NRS), with a lower score representing less disease activity.
Time Frame: At baseline and week 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion
Number analyzed (Participants) | 31 | 17
score on a scale
  Baseline: number analyzed (Participants) | 28 | 17
  Baseline | 7.1 (2.1) | 7.1 (2.1)
  Week 13: number analyzed (Participants) | 23 | 13
  Week 13 | 6.2 (2.3) | 5.4 (2.8)

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety criterion
Time Frame: Through study completion, up to Week 28
Measure: Count of Participants; unit: Participants
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion
Number analyzed (Participants) | 31 | 17
Participants
  Patients having reported at least one treatment emergent adverse event (TEAE) | 24 | 11
  Patients having reported at least one serious AE | 3 | 1

ADVERSE EVENTS:
Time Frame: Through Week 28 (about 6 months)
Arm/Group | S95011 Concentrate for Solution for Infusion | S95011 Placebo Concentrate for Solution for Infusion
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/17
Serious Adverse Events (participants affected / at risk) | 3/31 | 1/17
Other Adverse Events (participants affected / at risk) | 24/31 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S95011 Concentrate for Solution for Infusion (N=31) | S95011 Placebo Concentrate for Solution for Infusion (N=17)
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S95011 Concentrate for Solution for Infusion (N=31) | S95011 Placebo Concentrate for Solution for Infusion (N=17)
COVID-19 (Infections and infestations) | 5 | 2
Parotitis (Infections and infestations) | 2 | 1
Oral Herpes (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Salivary gland pain (Gastrointestinal disorders) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Discomfort (General disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT04605978/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT04605978/SAP_001.pdf